CLINICAL TRIAL: NCT01473485
Title: A Study to Evaluate the Safety and Feasibility of Transcranial MRI-Guided Focused Ultrasound Surgery in the Treatment of Brain Tumors
Brief Title: ExAblate (Magnetic Resonance-guided Focused Ultrasound Surgery) Treatment of Brain Tumors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT003
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Glioma; Metastatic Brain Cancer
Keywords: Brain Tumor; Glioma; Brain Cancer; Metastatic Brain Cancer
MeSH Terms: conditions — Glioma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ExAblate Transcranial Device (Experimental)
  Interventions: Device: ExAblate Transcranial System

INTERVENTIONS:
Device: ExAblate Transcranial System — MR Guided Focused Ultrasound
  Other Names: MRgFUS; FUS; Focused Ultrasound; MR Guided Focused Ultrasound

SUMMARY:
A Study to Evaluate the Safety and Feasibility of Transcranial MRI-Guided Focused Ultrasound Surgery in the Treatment of Brain Tumors

DETAILED DESCRIPTION:
Although the initial treatment of malignant gliomas is well established, the best treatment for progressive disease remains undefined. Patients with newly diagnosed gliomas are typically treated with surgery followed by conformal radiation and concomitant chemotherapy. Even though these tumors are not curable, prolonged survival can be achieved in selected patients. Despite improved multimodal therapies, almost all of the patients experience recurrence at the site of the primary tumor where they have already received maximal surgical resection and radiation therapy. Typically, these patients have a life expectancy of approximately 6 months, with less than a third of patients alive at one year. Salvage therapy for these patients usually take the form of various systemic chemotherapeutic agents because localized therapies such as reirradiation may not be possible in the previously irradiated site. As progressive disease has very poor response rates to current systemic therapies, efforts to define the role of novel local therapies, such as MR guided focused ultrasound (MRgFUS), is necessary.

There are very few local therapy options for progressive gliomas. Traditionally, reirradiation and surgery are considered last resort treatments for symptomatic recurrence. In the initial treatment of gliomas, the tumor and surrounding brain receive near tolerance doses and usually preclude a second course of radiation therapy. If clinically advisable and feasible, a second operation may be undertaken but is usually reserved for younger patients with a good neurological status who are developing neurological symptoms related to the mass effect of the tumor. The use of MR guided focused ultrasound represents a new, noninvasive therapeutic option that overcomes some of the limitations of secondary surgery or reirradiation and provides the patient with an option for local ablative therapy. The lesioning of the tumor is done accurately under MRI guidance with real-time monitoring of the ablative ultrasonic hyperthermia. As the cytotoxic affects are due to hyperthermia, there is no cumulative radiation affect which limits the use of radiotherapy in recurrent disease. The potential benefits for the patient include local control of the disease/tumor, and prolonging the time to subsequent salvage therapies.

A similar situation exists for brain metastases. Historically, the development of brain metastases was considered a terminal event, however, with better local therapies as well a systemic therapies, patients are living longer. Initial management of patients with brain metastases usually involves surgery, whole brain radiation, radiosurgery or a combination of these modalities depending on the clinical situation. The goal of treating brain metastases is to prevent the patient from succumbing to CNS disease. As improved systemic therapy has lengthened the survival of patients with metastatic tumors, more patients are surviving and developing recurrent or progressive metastatic CNS disease. Progressive disease usually requires more local therapies as chemotherapeutic agents do not adequately cross the blood brain barrier to have a large impact on CNS metastases. MRIgFUS could play and important role in ablating brain metastases in patients who have already been maximally radiated and are otherwise without options.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women.
2. Age between 18 and 75 years, inclusive.
3. Able and willing to give informed consent.
4. Able to tolerate pre / post - procedure steroid treatment
5. Subjects with recurrent or progressive glioma who have failed standard therapy with surgery and/or radiation for whom local therapy has been requested by the neuro-oncologist. This treatment will be offered as an option for those patients where neither surgery or repeat radiotherapy is advised by the multidisciplinary team.

   OR Patients with metastatic brain cancer that has progressed despite prior radiotherapy and local therapy is requested by the oncologist. This treatment will be offered as an option for those patients where surgery is not indicated and discussed with the potential options for repeat radiotherapy or salvage radiosurgery by the multidisciplinary team.
6. The targeted tumor tissue is located in the cerebral hemispheres, > 2.5 cm from the inner table of the skull. Non-targeted parts of the tumor may extend outside the treated tumor limits.
7. Tumor(s) are clearly defined on pre-therapy contrast enhanced MRI scans.

   * No more than 1 Brain Met can be treated under this protocol
8. Size of the targeted portion of the tumor (i.e. prescribed ROT) is less than 2.5 cm in diameter (8 cm3 in volume). The non-targeted tumor tissue may exceed the targeted volume.
9. Karnofsky rating 70-100.
10. ASA score 1-3.
11. Able to communicate sensations during the ExAblate MRGFUS procedure.
12. Able to attend all study visits (i.e., life expectancy of at least 3 months).
13. At least 14 days passed since last brain surgery or radiation therapy.

Exclusion Criteria:

1. The tumor's not visible on the pre-therapy imaging
2. The tumor presenting the following imaging characteristics

   * Brain edema and/or mass effect that causes midline shift or shift in wall of the third (3rd) ventricle of more than 10-mm.
   * Targeted area (i.e.: ROT) less than 5 millimeters from primary branches of cerebral vessels, dural sinuses, the hypophysis or cranial nerves
   * Evidence of recent (less than 2 weeks) intracranial hemorrhage.
   * Containing calcifications in the focused ultrasound sonication beam path in the event system tools cannot tailor the treatment around these calcification spots
3. The sonication pathway to the tumor involves

   * More than 30% of the skull area traversed by the sonication pathway is covered by scars, scalp disorders (e.g., eczema), or atrophy of the scalp.
   * Clips or other metallic implanted objects in the skull or the brain, except shunts.
4. The subject presents with:

   * Symptoms and signs of increased intracranial pressure (e.g., headache, nausea, vomiting, lethargy, and papilledema).
   * Unstable hemodynamic status including:
   * Documented myocardial infarction within six months of enrollment.
   * Symptomatic coronary artery stenosis.
   * Congestive heart disease not controlled by medication.
   * Cardiac pacemaker.
   * Severe hypertension (diastolic BP > 100 on medication).
5. Anti-coagulant therapy, on medications known to increase risk of hemorrhage, (e.g.: non-steroidal anti-inflammatory drugs (NSAIDs), statins)
6. Patients with history of bleeding disorder or with history of spontaneous haemorrhage tumour
7. Abnormal level of platelets (< 100000), PT (>14) or PTT (>36), and INR > 1.3.
8. Documented cerebral infarction within past 12 months
9. TIA or stroke in the last 1 month.
10. Patients with cerebral or systemic vasculopathy:

    * Symptomatic systemic vascular disease is defined as cardiovascular disease which prevents any procedure in MRI where ECG cannot be obtained (i.e. coronary disease). These patients must be excluded
11. Insulin-dependent diabetes mellitus.
12. Patients taking immunosuppressants (corticosteroids to prevent/treat brain edema are permitted).
13. Known sensitivity to gadolinium-DTPA.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-04; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate Safety of ExAblate Transcranial Device | At the time of ExAblate procedure
  To evaluate the incidence and severity of Adverse Events (AEs) associated with the ExAblate Transcrainal device during ExAblate treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada